CLINICAL TRIAL: NCT05120570
Title: PTCy + Sirolimus/VIC-1911 as GVHD Prophylaxis in Myeloablative PBSC Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021LS006; MT2021-01 (Other: University of Minnesota)
Record Dates: First submitted 2021-11-03; First posted 2021-11-15 (Actual); Results first posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Acute Leukemia; Myelodysplastic Syndromes; Myeloproliferative Neoplasm; Lymphoma
Keywords: VIC-1911; PTCy; Myeloablative; Allogeneic
MeSH Terms: conditions — Myelodysplastic Syndromes; Myeloproliferative Disorders; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PTCy/sirolimus plus VIC-1911 (Experimental): Patients enrolled and treated with PTCy/sirolimus plus VIC-1911
  Interventions: Drug: VIC- 1911

INTERVENTIONS:
Drug: VIC- 1911 — 25 mg, 50 mg, or 75 mg administered twice a day from day 5 post HCT to day 45, and the dose escalation will stop once we identify the lowest biologically active and safe dose of VIC.

SUMMARY:
This is a single-arm, phase I/II, study of PTCy/sirolimus plus VIC-1911 to prevent GVHD and relapse after Allogeneic Hematopoietic Cell Transplantation (alloHCT).

DETAILED DESCRIPTION:
Determination of the optimal dose during the Phase I trial is based on Dose Limiting Toxicity for safety and reduction of CD4+, pH3ser10+ T cells (phosphorylated histone 3 serine 10 is a biomarker of Aurora kinase A activity) for efficacy. Phase II will be powered to improve grade III-IV acute graft-versus-host disease and relapse after alloHCT, compared to historical estimates at the University of Minnesota.

Patients will receive myeloablative conditioning (MAC) with total body irradiation (TBI) followed by infusion of HLA-matched related or unrelated peripheral blood stem cells (PBSC) on day 0. Cyclophosphamide will be administered on days +3 and +4. Sirolimus targeting 8-12ng/ml will begin on day +5 until day +365. VIC-1911 will be administered as 25 mg, 50 mg, or 75 mg orally BID from day +5 to day +45 according to the rules of our phase I study. The lowest biologically active and safe dose of VIC-1911 will be identified as the recommended phase II dose.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of

  * acute leukemia in complete remission, or
  * myelodysplasia with <5% blasts, or
  * myeloproliferative neoplasm/myelofibrosis with <5% marrow or circulating blasts
  * chemosensitive Hodgkin or non-Hodgkin lymphoma
* Age 18 years or older
* Performance status of ≥ 80% Karnofsky
* Adequate organ function within 28 days of study registration defined as:

  * left ventricular ejection fraction ≥ 45%
  * pulmonary function with FEV1, FVC, and DLCO ≥ 50% predicted
  * AST and ALT < 2 times upper limit of normal
  * Total bilirubin <1.5 times the upper limit of normal. If the patient is suspected of having Gilbert syndrome, they require prior approval of the medical monitor
  * creatinine clearance ≥ 50cc/min
  * no active/uncontrolled infection
  * negative HIV, HBV and HCV
  * ferritin < 2000 ng/ml
* Patients able to tolerate oral medication
* Women of childbearing potential and men with partners of child-bearing potential must agree to use of contraception for the duration of treatment through 60 days after the last treatment of VIC-1911 or sirolimus
* Able to provide written voluntary consent prior to the performance of any research related tests or procedures

Exclusion Criteria:

* HCT-CI > 4 or unable to receive myeloablative TBI
* Use of planned post-transplant maintenance therapy to begin prior to day +75. Patients may receive standard of care maintenance therapies starting at day

  +75 or later
* Patients with a history of hypersensitivity to any of the investigational products
* Pregnant or breastfeeding as agents used in this study are Pregnancy Category

  o C: Drugs which, owing to their pharmacological effects, have caused or may be suspected of causing, harmful effects on the human fetus or neonate without causing malformations, and Pregnancy category D: There is positive evidence of human fetal risk based on adverse reaction data from investigational or marketing experience or studies in humans, but potential benefits may warrant use of the drug in pregnant women despite potential risks. Females of childbearing potential must have a negative pregnancy test (serum or urine) within 28 days of study registration.
* Women or men of childbearing potential unwilling to take adequate precautions to avoid unintended pregnancy from the start of protocol treatment through 60 days after the last treatment of VIC-1911 or sirolimus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2025-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherman Holtan, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were enrolled into the Phase II portion of the study. We concluded the trial when Phase Ia was completed, rather than proceeding to Phase Ib, due to funding constraints and the goal of focusing on developing a new randomized study.
Groups:
- Dose Level A1: 25 mg administered twice a day from day 5 post HCT to day 45. Dose escalation will stop once we identify the lowest biologically active and safe dose of VIC.
- Dose Level A2: 50 mg administered twice a day from day 5 post HCT to day 45. Dose escalation will stop once we identify the lowest biologically active and safe dose of VIC.
- Dose Level A3: 75 mg administered twice a day from day 5 post HCT to day 45. Dose escalation will stop once we identify the lowest biologically active and safe dose of VIC.
Period: Overall Study
Arm/Group | Dose Level A1 | Dose Level A2 | Dose Level A3
Started | 4 | 3 | 9
Completed | 3 | 3 | 9
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level A1 | Dose Level A2 | Dose Level A3 | Total
Number analyzed (Participants) | 4 | 3 | 9 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 8 | 15
  >=65 years | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 4 | 6
  Male | 4 | 1 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 3 | 9 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 4 | 1 | 8 | 13
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Determine the Optimal Dose of VIC-1911 When Given in Combination With Standard Immunosuppressive Therapy in Adult Patients Undergoing Myeloablative Stem Cell Transplantation.
Description: The optimal dose will be identified using the EffTox design. The proportion of patients with an average CD4+, pH3ser10+ T cell of <54%. The minimum desired biologic efficacy is 65% of patients by day 21 (+/- 3 days) with <30% of patients experiencing a DLT. Data only to reported from arm with maximum tolerated dose.
Time Frame: 21 days post treatment
Measure: Number; unit: mg of VIC
Arm/Group | PTCy/Sirolimus Plus VIC-1911
Number analyzed (Participants) | 15
mg of VIC | 75

2. Primary Outcome: Progression-free Survival
Description: Participant progression-free survival assessed using aGVHD data.
Time Frame: 1 Year
Measure: Number; unit: Percentage of participants
Arm/Group | Dose Level A1 | Dose Level A2 | Dose Level A3
Number analyzed (Participants) | 3 | 3 | 9
Percentage of participants | 100 | 100 | 100

3. Primary Outcome: Relapsed Assessment (Phase I)
Description: Assessment to determine if patient has relapse in MTD arm. Data only to reported from arm with maximum tolerated dose.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dose Level A3
Number analyzed (Participants) | 9
Percentage of participants | 0 [0 to 0]

4. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival for participants on MTD arm. Data only to reported from arm with maximum tolerated dose.
Time Frame: 1 year
Measure: Number; unit: Percent of participants
Arm/Group | Dose Level A3
Number analyzed (Participants) | 9
Percent of participants | 100

5. Secondary Outcome: To Determine the Cumulative Incidences of Acute GVHD
Description: Assessment of aGVHD for MTD arm. Data only to reported from arm with maximum tolerated dose.
Time Frame: Day 100
Measure: Number (95% Confidence Interval); unit: number of new cases per 900 person-days
Arm/Group | Dose Level A3
Number analyzed (Participants) | 9
number of new cases per 900 person-days | 6 [2 to 10]

6. Secondary Outcome: To Determine the Cumulative Incidences of Chronic GVHD
Description: Assessment of cGVHD
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dose Level A1 | Dose Level A2 | Dose Level A3
Number analyzed (Participants) | 3 | 3 | 9
Percentage of participants | 0 [0 to 0] | 0 [0 to 0] | 33 [4 to 63]

7. Secondary Outcome: Progression-free Survival Comparing Graft-Versus-Host Disease-Free (GRFS) to the Standard PTCY Plus Tacrolimus/Mycophenolate Mofetil Regimen From MT2015-29
Description: Progression-free Survival assessed using GRFS defined as grade III-IV acute GVHD, chronic GVHD requiring immunosuppression, relapse, or death by 1 year
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dose Level A1 | Dose Level A2 | Dose Level A3
Number analyzed (Participants) | 3 | 3 | 9
Percentage of participants | 100 [0 to 100] | 100 [0 to 100] | 67 [28 to 88]

8. Secondary Outcome: Progression Free Survival
Description: Percentage of participants with progression free survival at 1 year for MTD arm. Data only to reported from arm with maximum tolerated dose.
Time Frame: 1 Year
Measure: Number; unit: Percent of participants
Arm/Group | Dose Level A3
Number analyzed (Participants) | 9
Percent of participants | 100

9. Secondary Outcome: Frequency of CMV Reactivation and Disease
Description: Analyze the frequency of CMV reactivation and disease for MTD arm. Data only to reported from arm with maximum tolerated dose.
Time Frame: Day 100
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dose Level A3
Number analyzed (Participants) | 9
Percentage of participants | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Dose Level A1 | Dose Level A2 | Dose Level A3
All-Cause Mortality (participants affected / at risk) | 1/4 | 0/3 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/4 | 2/3 | 3/9
Other Adverse Events (participants affected / at risk) | 1/4 | 3/3 | 3/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level A1 (N=4) | Dose Level A2 (N=3) | Dose Level A3 (N=9)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (4)
Skin and subcutaneous tissue disorders - Other, specify - Sweet's syndrome (acute febrile neutro (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, specify - Histoplasmosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Immune system disorders - Other, specify - Immune Reconstitution Inflammatory Syndrome. (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Vascular disorders, hematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level A1 (N=4) | Dose Level A2 (N=3) | Dose Level A3 (N=9)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Keratitis (Eye disorders) | 0 (0) | 3 (3) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Histoplasmosis) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (skin lesions) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Sweet's syndrome) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Vascular disorders - Other, specify (hematoma) (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-08): https://cdn.clinicaltrials.gov/large-docs/70/NCT05120570/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-08): https://cdn.clinicaltrials.gov/large-docs/70/NCT05120570/ICF_001.pdf